CLINICAL TRIAL: NCT06225661
Title: Focused Suicide Prevention Strategy for Youth Presenting to the Emergency Department With Suicide Related Behaviour: A Multi-site Randomized Controlled Trial
Brief Title: Focused Suicide Prevention Strategy for Youth Presenting to the Emergency Department With Suicide Related Behaviour
Acronym: IAMSAFE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); SickKids Foundation (Other)
Responsible Party: Principal Investigator, Daphne Korczak, Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB1000056892
Record Dates: First submitted 2024-01-11; First posted 2024-01-26 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Suicide; Suicide Prevention; Suicidal Ideation; Self-Injurious Behavior; Behavioral Symptoms; Suicide, Attempted; Suicide and Self-harm
MeSH Terms: conditions — Suicide; Suicide Prevention; Suicidal Ideation; Self-Injurious Behavior; Behavioral Symptoms; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study investigators and outcome assessors are blinded to allocation assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAFE Intervention (Experimental): This group will receive the SAFE individual youth and family-based intervention.
  Interventions: Behavioral: SAFE Intervention
- NAV (Telephone Navigation) (Active Comparator): This group will receive telephone-based case navigation.
  Interventions: Behavioral: NAV (Telephone Navigation)

INTERVENTIONS:
Behavioral: SAFE Intervention — Manualized individual youth and family psychotherapeutic intervention. Weekly individual and family sessions with a therapist for 6 weeks. Participants will continue to receive usual care.
  Arms: SAFE Intervention
Behavioral: NAV (Telephone Navigation) — Weekly telephone contact with parents regarding participant health care utilization. Referrals to community mental health resources provided as needed. Participants will continue to receive usual care.
  Arms: NAV (Telephone Navigation)

SUMMARY:
Suicide is the leading cause of death due to illness among Canadian youth, claiming more lives than any medical illness, including cancer. Suicide prevention is possible, and early intervention is needed. The investigators will examine the effectiveness of a previously-piloted, ED-based suicide prevention intervention, across Canadian sites, using a randomized clinical trial design. The investigators will determine whether the patient- and family-centered intervention is more effective than enhanced usual care in reducing suicide-related behaviors in 330 youth at high-risk of suicide.

DETAILED DESCRIPTION:
This is a Multi-site Randomized Controlled Trial of a patient- and family-centered suicide prevention intervention added to usual care (SAFE + UC) for adolescents aged 12 to 17 years who present to the Emergency Department (ED) with suicidal ideation or suicide risk behaviours. The investigators will determine whether the SAFE + UC intervention is more effective than enhanced usual care (telephone navigation + UC) in reducing suicide-related behaviors in 330 youth at high-risk of suicide across Canadian sites.

SAFE + UC is a 6-week, standardized, manualized outpatient program that teaches participants to the skills to manage suicidal thoughts and impulses effectively. The family component addresses conflictual relationships that may be present in the family as well as improving family communication.

Telephone navigation (NAV) + UC consists of up to 6 weekly telephone calls to ensure that the participant has connected with community resources suggested by the ED team and provide additional resources as needed.

ELIGIBILITY:
Inclusion Criteria:

* Youth presenting in the Emergency Department with SIQ-Jr score ≥ 31,
* Has a participating parent or caregiver who is able to communicate easily in English, or is willing to communicate using a hospital-organized translator,
* Between the ages 12-17 years old,
* Living in the catchment area of one of the three hospital sites and access to a telephone.

Exclusion Criteria:

* Score of 3 on KSADS screen for current psychosis or elevated mood
* Moderate to severe intellectual disability, and/or autism based on clinical chart.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Suicide Risk Events (SREs) throughout 6 months of study engagement | Baseline, 6 weeks, 24 weeks
  Suicide attempts and unscheduled ED/hospital re-visits (including hospitalization) for SREs, or death by suicide during the 6-month follow up period. SREs will be determined by participant and caregiver report using validated questions regarding suicide attempts from the Columbia-Suicide Severity Rating Scale (C-SSRS).

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, 6 weeks, 24 weeks
  The Columbia-Suicide Severity Rating Scale is an interviewer-administered measure used to assess intensity of suicidal ideation and severity of suicidal behavior. Questions 1-5 (Ideation Severity Subscale) gage five types of ideation of increasing severity, scoring presence/absence of any suicidal ideation yes or no. The most severe ideation endorsed (1-5) becomes the score for this section. The Intensity of Ideation Subscale sums 5 items endorsed. Sums range from 2 to 25, with higher scores indicating more intense ideation. The Suicidal Behavior Subscale scores 4 types of suicidal behaviors; yes or no and identify categorical occurrence and density of actual, interrupted, aborted attempts and preparatory behaviors and distinguish suicidal and non-suicidal self injurious behavior.
Suicidal Ideation Questionnaire-Jr (SIQ-Jr) | Baseline, 6 weeks, 24 weeks
  The Suicidal Ideation Questionnaire-Jr (SIQ-Jr) measures intensity of suicidal ideation. The SIQ-Jr is a 15-item self-report questionnaire that assesses suicidal thoughts on a 7-point scale. Scores range from 0 to 90, with higher scores indicative of more severe suicidal ideation.
Schedule for Affective Disorders and Schizophrenia Depression Rating Scale (KSADS-DEPc) | Baseline, 6 weeks, 24 weeks
  Semi-structured interviewer-administered diagnostic measure designed for use with children and adolescents. Youth are asked about past month depression symptoms and suicidality to determine the presence or absence of a diagnosis of depression.
Screen for Child Anxiety Related Disorders (SCARED) | Baseline, 6 weeks, 24 weeks
  Measure of youth anxiety symptoms by self-report. There are 41 items in the measure. Scores range from 0-82, with higher values indicating greater anxiety symptoms.
Centre for Epidemiological Studies Depression Scale for Children (CES-DC) | Baseline, 6 weeks, 24 weeks
  Measure of youth depressive symptoms by self-report. There are 20 items in the measure. Total scores range from 0-60, with higher values indicating greater depressive symptoms.
Life Problems Inventory (LPI) | Baseline, 6 weeks, 24 weeks
  Measure of four core problem areas of borderline personality disorder by youth self-report. There are 60 items in the measure. Scores range from 60-300, with higher values indicating worse symptoms.
Columbia Impairment Scale (CIS) | Baseline, 6 weeks, 24 weeks
  Measure to assess global functioning and impairment by self- and parent- report. There are 13 items in the measure. Scores range from 0-52, with higher scores indicating greater impairment.
Conflict Behaviour Questionnaire (CBQ) | Baseline, 6 weeks, 24 weeks
  The CBQ is a 20-item self- and parent-report instrument that assesses aspects of the parent-child relationship including communication and conflict within the relationship. One measure is completed for each specific child-parent relationship. Scores range from 0-20, with higher scores indicating greater conflict.
Cost-Effectiveness Ratio | Baseline, 6 weeks, 24 weeks
  Cost effectiveness will be expressed as the incremental cost-effectiveness ratio, calculated by dividing the incremental costs between study arms by the incremental change in SREs per participant between baseline and 6 months. Data regarding directs and indirect costs incurred by youth and caregivers will be collected using an interviewer-administered survey developed by the study team. Cost-effectiveness will be determined as funding allows. Direct costs (intervention, medication, health services use) will be collected from investigators and participants. Indirect costs will include out-of-pocket expenses and productivity losses experienced by participants and their caregivers
Treatment Fidelity (Adherence and Competence) to the SAFE Intervention | Baseline, 6 weeks, 24 weeks
  Adherence to the core components of the intervention will be assessed using the Fidelity Treatment Checklist, a 10-item independent rater- and therapist-rated measure developed for the SAFE intervention based on existing measures of individual therapy and family therapy implementation fidelity. Scores range from 0-20, with higher scores indicating greater fidelity.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Alberta Children's Hospital - Alberta Health Services & University of Calgary, Calgary, Alberta
  - McMaster Children's Hospital - Hamilton Health Sciences, Hamilton, Ontario
  - Trillium Health Partners, Mississauga, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No